CLINICAL TRIAL: NCT07254481
Title: A Phase 1, Randomized, Double-Blind Placebo-Controlled Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, Food Effects, and QT/QTc Interval Impact of VB19055 Tablets in Healthy Chinese Adult Subjects
Brief Title: VB19055 Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in a Healthy Chinese Population
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Yangli Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB19055-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Doses (SAD, Part A) (Experimental): In this part, 5 ascending dose cohorts (8 participants per cohort) will be studied. Within each cohort, participants will be randomized in a 3:1 ratio to receive either VB19055 or placebo.
  Interventions: Drug: VB19055; Drug: VB19055 placebo
- Food Effect (FE, Part B) (Experimental): 14 participants and single dose food effect cohort. This part is open-label, two sequence, two-period, crossover design.
  Interventions: Drug: VB19055
- Single Ascending Doses (MAD,Part C) (Experimental): In this part, 4 ascending dose cohorts (8 participants per cohort) will be studied. Within each cohort, participants will be randomized in an 3:1ratio to receive either VB19055 or placebo.
  Interventions: Drug: VB19055; Drug: VB19055 placebo

INTERVENTIONS:
Drug: VB19055 — In this part, VB19055 tablets will be administered as a single or multiple oral dose.
Drug: VB19055 placebo — In this part, VB19055 placebo tablets will be administered as a single or multiple oral dose.
  Arms: Single Ascending Doses (MAD,Part C); Single Ascending Doses (SAD, Part A)

SUMMARY:
The purpose of this study is to evaluate the safety,tolerability,pharmacokinetics and pharmacodynamics of VB19055 in the healthy Chinese population.

DETAILED DESCRIPTION:
This trial contains Part A, Part B and Part C, all enrolling healthy Chinese subjects.

Part A is a single ascending dose study of VB19055 tablets in healthy Chinese adult participants. Part B is a randomized, single-dose, two-period, crossover study designed to evaluate the effect of food on the pharmacokinetic characteristics of VB19055 tablets in healthy Chinese adult participants.Part C is a multiple ascending dose study of VB19055 tablets in healthy Chinese adult participants.

Part A will be conducted first, and Parts B and C will be initiated when appropriate based on the preliminary data obtained during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical trials, understand the nature of the study and any risks involved in participation, sign an informed consent form, and be willing to comply with the requirements specified in the protocol;
2. Aged between 18 and 50 years (inclusive), healthy volunteers;
3. Body mass index (BMI) between 18-26 kg/m² (inclusive), with minimum weight requirements of 50 kg (inclusive) for males and 45 kg (inclusive) for females;
4. In generally good health, as determined by the investigator based on medical history, surgical history, complete physical examination, vital signs measurements, laboratory tests, 12-lead electrocardiogram (ECG), and chest X-ray results, with no evidence of clinical disease and confirmed to be healthy;
5. For females of childbearing potential: Agree to use highly effective contraception (e.g., intrauterine device, hormonal contraceptives, or condoms) throughout the study and for 3 months after the last dose, with a negative serum pregnancy test at screening.

For males: Agree to use effective contraception (specific methods detailed in Appendix 5) during the study and for 3 months after the last dose.

Exclusion Criteria:

1. Known allergy to aldosterone synthase inhibitors or any components/excipients of the investigational drug;
2. The clinically significant endocrine, metabolic, cardiovascular, respiratory, gastrointestinal, liver and kidney, nervous system (including the history of seizures) or any significant history of mental illness or mental disorder, or clinically significant diseases, conditions or other evidence, which the researcher believes will pose risks to the safety of the subjects or interfere with the development, conduct or completion of the study;
3. Any known diseases or conditions that may interfere with drug absorption, distribution, metabolism or excretion (such as dysphagia or gastrointestinal diseases that affect drug absorption, or previous gastric surgery, vagotomy, enterotomy or any surgery that may interfere with gastrointestinal peristalsis, PH or absorption, etc.);
4. Vaccination with active or attenuated vaccine within 4 weeks before screening or during the trial (except influenza vaccine);
5. Drinking excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250mL) per day, or drinking tea, coffee and/or caffeinated beverages within 48 hours before drug administration, or unable to stop drinking during the trial; Had a history of long-term consumption of a beverage or food rich in xanthine or grapefruit, or had taken any product rich in xanthine or grapefruit within 48 hours before administration；
6. Smokers or those who used nicotine products excessively (≥5 cigarettes per day on average) in the 3 months before screening or who were unable to stop using any tobacco or nicotine-based products (snus, chewing tobacco, cigars, pipes, or nicotine-replacement products) during the trial；
7. Participants who had participated in a clinical trial of another drug and had taken any investigational drug within 3 months before the first dose；
8. Use of corticosteroids within 3 months prior to the first dose；
9. Within 3 months before the first dose of blood donation or blood loss≥400 ml, blood transfusion or use of blood products, or plans to test during or within 30 days after the last drug blood donors；
10. Were heavy drinkers or regular drinkers in the 3 months before screening, which was defined as having consumed an average of 14 standard units of alcohol per week (one unit of alcohol =285mL of beer or 25mL of spirits or 125mL of wine), had a positive alcohol breath test at screening, or were unable to stop using any alcohol-containing product during the trial;
11. Drug abuse screening is positive or in the past five years has a history of substance abuse or screening before 3 months used drugs；
12. Blood pressure in the range of 90-140mmHg (systolic) or 50-90mmHg (diastolic) or pulse rate in the range of 50-100 beats/min during the screening period;Or postural hypotension (systolic blood pressure decreased ≥20mmHg or diastolic blood pressure decreased ≥ 10mmHg while standing)；
13. During the screening period, any one of the infectious disease screening results of hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibody, HIV antibody and treponema pallidum antibody was positive；
14. The presence of uncontrolled active bacterial, viral, fungal, rickettsial, or parasitic infections, unless treated prior to study treatment and had returned to normal；
15. Use of any medication (including prescription drugs, over-the-counter drugs, herbal medicines, functional vitamins, supplements, etc.) within 14 days before the first dose (or within 5 half-lives of the drug used, whichever is longer) that the investigator considers may affect the evaluation of the pharmacokinetic characteristics of the study drug or interfere with the study procedures or affect the safety assessment；
16. Serum potassium level <3.5 mmol/L or ≥5.0 mmol/L at screening and admission；
17. Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin >1.5 times the upper limit of normal (ULN) at screening or admission；
18. Abnormal renal function (estimated glomerular filtration rate < 90 mL/ minute /1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation, as described in Appendix 1: CKD-EPI equation)；
19. Family history of long or short QT syndrome, history of syncope or torsdes pointes, heart failure, or clinically significant/symptomatic bradycardia, and risk factors including uncontrolled hypokalemia, hypocalcemia, or hypomagnesemia.For participants in the QT/QTc study, use of antiarrhythmic drugs, inotropic drugs, beta-blockers, calcium-channel blockers, quinolones, and other drugs with a risk of prolonging the QT/QTc interval or causing torsdes pointes within 4 weeks before the first dose (see Appendix 3 for details); And prolonged QTcF interval (> 450msec)；
20. Clinically significant abnormal ECG findings at screening or admission as judged by the investigator; Strenuous physical training or excessive exercise (e.g., long-distance running, weight lifting, or any physical activity to which the participant is not accustomed) from 7 days before administration until the end of the study；
21. The investigator judged that the subject had other conditions that were not suitable for participation in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events as assessed by CTCAE v5.0 | Average half a month
  The rate of Adverse events occur during the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Hangzhou First People's Hospital, Hangzhou
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No